CLINICAL TRIAL: NCT07124832
Title: A Pragmatic Randomized Controlled Pilot Trial for Weight Loss in Patients With Obesity: Assessment of the Socratic Questioning Method
Brief Title: Intervention Study on Weight Loss in Patients With Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sıdıka Ece Yokuş (Other)
Responsible Party: Sponsor-Investigator, Sıdıka Ece Yokuş, Research Assistant, Celal Bayar University
Organization: Celal Bayar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20.478.486/3150
Record Dates: First submitted 2025-08-06; First posted 2025-08-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to intervention and control groups at a 1:1 ratio using the block randomization method (block size 6) with a computer-aided program.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socratic Questioning Group (Active Comparator): Participants in the intervention group will be followed up by physicians using the Socratic questioning technique. Face-to-face meetings will be held on the 0th, 15th, 30th and 60th days, and each session will take approximately 10-15 minutes. Physicians will use a checklist and ICD-10 code (E66: Obesity) when recording participant notes. The group to which the participant is assigned will be indicated in the Family Medicine Information System, and this warning note will be visible to physicians at each examination. Researchers will not interfere with the content of the interview, and physicians will be given flexibility to apply the Socratic questioning technique according to the needs of the participant.
  Interventions: Behavioral: Socratic Questioning Method
- Regular Care Group (No Intervention): Participants in the control group will be followed up with the routine obesity approach used by physicians in their daily practice. Physicians will maintain the standard of care they normally give to patients with obesity. This approach may include nutritional advice, physical activity recommendations, and general lifestyle change advice, but Socratic questioning techniques will not be used.

INTERVENTIONS:
Behavioral: Socratic Questioning Method — Socratic questioning is a method in which behaviour is examined through questions such as "what, where, which, who, when, how, and why". It consists of four stages: defining the problem, evaluating and identifying alternatives, redefining, and discussing feasible outcomes. Through this process, individuals develop their critical thinking skills and make self-evaluations.
  Arms: Socratic Questioning Group

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of using Socratic questioning as an alternative method for weight loss in adult patients with obesity (aged 18 to 65) in a primary care setting.

The main question it aims to answer is:

-Is Socratic questioning an effective alternative approach for promoting weight loss in patients with obesity?

Researchers will compare participants receiving Socratic questioning during follow-up visits with those receiving regular care to see if the intervention leads to greater weight loss.

Participants will:

* Complete a baseline questionnaire including 9 demographic questions and the 14-item Hospital Anxiety and Depression Scale (approx. 5 minutes).
* Attend five in-person follow-up visits with their family physician over a 3-month period (every 15 or 30 days), where they will receive brief counseling (10-15 minutes per visit) and have their weight, height, and waist circumference measured.
* Complete a 17-question final questionnaire at the end of 3 months (approx. 10-15 minutes).
* Be referred to mental health services if necessary, based on initial screening results.

DETAILED DESCRIPTION:
Work Packages:

1. Providing training to physicians on Socratic questioning:

   Training will be delivered online by an instructor experienced in cognitive behavioral therapy.
2. Recruitment of patients:

   During routine outpatient visits, physicians will assess patients diagnosed with obesity according to inclusion and exclusion criteria. Eligible patients will be recruited after providing informed consent. Patients will complete an information form and the Hospital Anxiety and Depression Scale (HADS). Those with significant psychopathology will be referred to a specialist for psychiatric evaluation. A first appointment (Day 0) will be scheduled.
3. Group allocation:

   After recruiting a patient, the physician will contact the research team to learn the patient's group assignment. The physician will be informed about the assigned group. Group allocation will be based on a pre-prepared list using computer-assisted block randomization.
4. Recording group assignment in the health information system:

   The patient's assigned group will be recorded in the Family Medicine Information System, and a reminder note will be visible during each consultation.
5. Physician-patient consultation on Day 0:

   The physician will take measurements and provide counseling about obesity. In the intervention group, the physician will apply the Socratic questioning technique. In the control group, the physician will follow routine obesity management practices. The next appointment (Day 15) will be scheduled.
6. Physician-patient consultation on Day 15:

   The physician will provide counseling about obesity. No measurements will be taken at this visit. The next appointment (Day 30) will be scheduled.
7. Physician-patient consultation on Day 30:

   The physician will provide counseling and take measurements. The next appointment (Day 60) will be scheduled.
8. Physician-patient consultation on Day 60:

   The physician will provide counseling and take measurements. The next appointment (Day 90) will be scheduled.
9. Physician-patient consultation on Day 90:

   Final measurements will be taken, and the study participation will be completed.
10. Data analysis:

    Physicians will share the collected data with the research team. The data from this pilot study will be analyzed.
11. Process evaluation:

At the end of the study, surveys including Likert-scale, multiple-choice, and open-ended questions will be administered to physicians and patients in the intervention group by the research team.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Body Mass Index (BMI) ≥ 30 kg/m²
* Willingness to participate in the study

Exclusion Criteria:

* Pregnancy or breastfeeding
* Presence of active psychosis or manic episode
* Intellectual disability
* Severe depression or personality disorder
* Auto- or hetero-aggressive behavior
* Reported use of psychoactive substances
* Suicidal ideation
* Participation in another weight loss program within the last 6 months
* Use of medications that cause long-term weight gain or loss
* Detection of psychopathology based on the Hospital Anxiety and Depression Scale (HADS)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Body Weight at 3 Months | Baseline and 3 months
  Body weight will be measured in kilograms using a calibrated digital scale. The outcome is the difference in percent change in body weight from baseline to 3 months between the Socratic questioning intervention group and the regular care control group.

SECONDARY OUTCOMES:
Change from Baseline in Body Mass Index (BMI) at 3 Months | Baseline and 3 months
  Body Mass Index will be measured in kg/m², calculated from weight (calibrated digital scale) and height (stadiometer). The outcome is the absolute change in BMI from baseline to 3 months.
Change from Baseline in Waist Circumference at 3 Months | Baseline and 3 months
  Waist circumference will be measured in centimeters using a non-elastic tape. The outcome is the absolute change in waist circumference (cm) from baseline to 3 months.
Association Between Weight Loss Percentage and Previous Attempts to Lose Weight | Baseline and 3 months
  Association between percentage weight loss from baseline to 3 months and self-reported previous weight loss attempts at baseline (yes/no).
Correlation Between Weight Loss Percentage and Baseline Willingness | Baseline and 3 months
  Correlation between percentage weight loss from baseline to 3 months and baseline willingness to create behavioral change score measured using a self-reported numerical rating scale (0-10, where 0=not willing at all and 10=extremely willing).

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Gómez Bravo, Study Director — Centre Hospitalier Neuro-Psychiatrique, Luxembourg; Vinicius Anjos de Almeida, Study Director — University of Sao Paulo; Sandra León Herrera, Study Director — University of Zaragoza, Spain; Sıdıka E. Yokuş, Principal Investigator — Manisa Celal Bayar University; Hüseyin Elbi, Study Director — Manisa Celal Bayar University
Locations (1):
- Manisa Celal Bayar University Mustafa Yardimci Education Family Health Center, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No data sharing plan was made due to the statement 'Your personal information will not be shared with any other person or organisation' in the ethics committee application file.